CLINICAL TRIAL: NCT04652856
Title: Neurocognitive Basis of Attention and Eye Movement Guidance in the Real World Scenes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We are withdrawing this study due to issues with recruitment. These issues arose as a result of the COVID-19 pandemic, effecting the availability of patients and our ability as a lab to work with these patients.
Sponsor: Avniel Ghuman (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor-Investigator, Avniel Ghuman, Associate Professor, Neurological Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY19090010; 1R21EY030297-01A1 (NIH)
Record Dates: First submitted 2020-11-04; First posted 2020-12-03 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Cognition; Attention; Eye Movements
Keywords: Visual Attention; Naturalistic Vision; Intracranial Electroencephalography; Electrical Brain Stimulation
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: All participants will undergo both electrical brain stimulation (EBS) and sham electrical brain stimulation (SEBS) at brain locations where alteration of visual attention behavior is expected to occur, as well as at control locations.
  The participants will be informed that they will receive both EBS and SEBS, but blinded to the location of each trial and whether the trial is EBS or SEBS. Participants will also be blinded to the objectives of stimulation.
  The order of stimulation locations and whether the trial is EBS or SEBS will be randomized.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Electrical and Sham Electrical Brain Stimulation (Experimental): Electrical brain stimulation and sham electrical brain stimulation will be administered to all participants.
  Interventions: Device: Electrical Brain Stimulation; Device: Sham Electrical Brain Stimulation

INTERVENTIONS:
Device: Electrical Brain Stimulation — Electrical Brain Stimulation (EBS) will be used to disrupt local neural activity in inferior temporal regions (ITC), parahippocampal cortex (PHC), the hippocampus, and control regions. The effects of EBS will be examined on attention and eye movement behavior, and all participants will receive both EBS and sham electrical brain stimulation.
Device: Sham Electrical Brain Stimulation — Sham electrical brain stimulation (SEBS) will be applied to inferior temporal regions (ITC), parahippocampal cortex (PHC), the hippocampus, and control regions. The effects of SEBS will be examined on attention and eye movement behavior, and all participants will receive both SEBS and EBS.

SUMMARY:
The objective of this study is to determine the effects of electrical brain stimulation (EBS) on visual search in natural scenes in humans.

DETAILED DESCRIPTION:
The ability to conduct a visual search for an object in a naturalistic scene is a crucial component of everyday interactions with the environment. This process requires the recognition of different items, accessing stored semantic knowledge about those items and their relationships with other objects, and guiding vision based on that knowledge. Classical models of attention emphasize low-level visual salience maps for attentional guidance. However, behavioral studies increasingly support a role for object knowledge in guiding attention and eye movements. Despite strong behavioral evidence that conceptual information about objects and scenes is critical for real world guidance of attention, very little is known about the neural basis of the guidance of attention based on meaning.

Previous human imaging studies have identified several brain regions that represent object and scene/context knowledge as it relates to visual recognition. In particular, regions of the temporal lobes (inferior temporal regions (ITC), parahippocampal cortex (PHC), and the hippocampus) are critical for perceiving and understanding objects, but little is known about the role of these individual regions in how they interact to guide attention and eye movements in real-world scenes.

Electrical brain stimulation is routinely performed clinically in the surgical treatment of epilepsy patients, both intraoperatively and using implanted electrodes. It is used as standard of care both to map eloquent brain function prior to surgical treatment for epilepsy and to map the seizure network. The purpose of this study is to gain a better understanding of the information flow and neural dynamics of the brain, examining the impact of electrical brain stimulation on stimulus search time, accuracy, and eye movement trajectories.

ELIGIBILITY:
Inclusion Criteria:

* Have intracranial EEG electrodes implanted for stage II epilepsy planning.
* Have adequate cognitive and communication ability to give informed consent, understand instructions, and follow direction.
* Be able to understand the tasks and provide responses.
* IQ > 75 (done as part of standard-of-care neuropsychological testing as part of the surgical treatment for epilepsy)
* Speak English

Exclusion Criteria:

* Inability to understand or perform the tasks outlined in this protocol
* In excessive postoperative discomfort.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of eye fixations during electrical brain stimulation (EBS) vs. sham electrical brain stimulation (SEBS). | Eye fixation incidence will be assessed during the intervention, through study completion, up to 1 week on average.
  Eye fixations will be assessed using an eye tracking device, which collects videos of eye movements. Participants will be presented with an image of a scene, and asked to locate a target object. The incidence of eye fixations occurring before participants locate the target object will be measured at preferred and control brain regions during EBS and SEBS.

SECONDARY OUTCOMES:
Search time for target object during EBS vs. SEBS. | Search Time will be assessed during the intervention, through study completion, up to 1 week on average.
  Visual search time will be assessed by asking participants to answer a simple question about a target object in an image of a scene as quickly and accurately as possible. The question will presented to the participants, followed by the image of the scene. The search time to locate the target object and respond to the question will be measured at preferred and control brain regions during EBS and SEBS.
Identification accuracy during EBS vs. SEBS. | Identification accuracy will be assessed during the intervention, through study completion, up to 1 week on average.
  Identification accuracy rate will be assessed based on the participants' correct responses for identifying a target object in an image of a scene (described in Outcomes 1 and 2). The search time to locate the target object will be measured at preferred and control brain regions during EBS and SEBS.

CONTACTS AND LOCATIONS:
Overall Officials: Avniel S Ghuman, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No